CLINICAL TRIAL: NCT06370923
Title: Harnessing Male Peer Networks to Enhance Engagement With HIV Prevention: A Large-scale Cluster Randomized Trial to Increase HIV Self-testing and PrEP Uptake Among Men in Eastern Zimbabwe
Brief Title: Harnessing Male Peer Networks to Enhance Engagement With HIV Prevention
Acronym: IMPERATIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: Biomedical Research and Training Institute, Zimbabwe (Other); Imperial College London (Other); University of Lincoln (Other); University College London Hospitals (Other); University of Copenhagen (Other); University of Washington (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, Frank Tanser, Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01MH133488-01 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-04-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
Keywords: HIV self test; HIV Pre Exposure Prophylaxis; Peer Networks
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial
Who Masked: Outcomes Assessor
Masking Description: Analysts blinded to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Distribution (Experimental): In intervention clusters investigators will identify initial distributors who will receive an HIVST kit for personal use and HIVST kits to distribute to local peers. These peers can subsequently become distributors, allowing the intervention to propagate through peer networks. A toll-free helpline will provide pre- and post-test support and an SMS-based risk assessment will expedite PrEP initiation at the clinic.
  Interventions: Behavioral: Peer Distribution
- Community Health Worker Distribution (Active Comparator): This will be the Standard of Care, HIVST kits distributed by Community health workers in the Control clusters.
  Interventions: Behavioral: Community Health Worker Distribution

INTERVENTIONS:
Behavioral: Peer Distribution — In intervention clusters investigators will identify initial distributors who will receive an HIVST kit for personal use and HIVST kits to distribute to local peers. These peers can subsequently become distributors, allowing the intervention to propagate through peer networks. A toll-free helpline will provide pre- and post-test support and an SMS-based risk assessment will expedite PrEP initiation at the clinic.
  Arms: Peer Distribution
Behavioral: Community Health Worker Distribution — Distribution of HIV self tests by community health workers
  Arms: Community Health Worker Distribution

SUMMARY:
Novel strategies are needed to engage men in Sub Saharan Africa (SSA) with HIV testing, treatment and prevention services to drive the epidemic towards elimination. Suboptimal engagement with HIV prevention by men increases their risk of HIV acquisition, and is an important driver of new HIV infections in women. HIV self-testing (HIVST) addresses several key facility-based access barriers and HIVST distribution through leveraging male peer networks for HIV prevention is feasible, acceptable and effective in SSA.

The objective of this project is to use an implementation science approach to establish the impact of HIVST distribution through male social networks, with phone-based support and improved risk perception, on PrEP (Pre-Exposure Prophylaxis) uptake among men in Eastern Zimbabwe. The project will leverage infrastructure and data associated with 20-year programme of HIV surveillance and behavioural research in a well-characterized population cohort hosted by the Manicaland Centre for Public Health Research, Zimbabwe.

The study will utilise a cluster randomised design of 44 clusters (22 Intervention:22 control) comprising on average 81 men in each cluster (total N = 3591) followed for 6 months (giving >80% power to detect a difference in PrEP initiation among men of 2% versus 8.5%). In intervention clusters the investigators will identify initial distributors who will receive an HIVST kit for personal use and HIVST kits to distribute to local peers. These peers can subsequently become distributors, allowing the intervention to propagate through peer networks. A toll-free helpline will provide pre- and post-test support and an SMS (Short Message Service) -based risk assessment will expedite PrEP initiation at the clinic. The study team will conduct a performance (process) evaluation of the intervention. to assess implementation fidelity, causal mechanisms underlying trial effectiveness including how characteristics of peer networks affect outcomes. Results of the study will be used to quantify the population level impacts and cost-effectiveness of male peer to peer HIVST distribution strategies on the uptake of PrEP in HIV hyper-endemic settings using a fully calibrated individual-based mathematical model. The envisaged long-term impact of this research is the development of a generalizable, multicomponent male peer-based HIVST and PrEP uptake model for settings where HIV incidence is high.

DETAILED DESCRIPTION:
The study will use a cluster-randomised trial design with clusters based on existing village boundaries, which have been utilised as part of an ongoing population-based HIV surveillance. In some cases, neighbouring villages will be aggregated to give approximately equal numbers of adult men in each cluster.

The study cohort from which participants will be recruited is located in Manicaland province, east Zimbabwe.

The intervention will proceed with the following steps:

i. Potential primary distributors will be identified by the research team following engagement with local key informants, these individuals will be contacted and screened for study enrolment. The desired characteristics of these individuals would be that they are members of their community with strong local networks of peers. If they choose to participate an informed consent procedure will be completed by the fieldworkers.

ii. If enrolled, the distributor will be given a pack containing four HIVST kits, one for their own use and three for distribution within the cluster. The study team will collect basic demographic data (name/age / cell number) for the distributor and the intended recipients. They will also record the unique ID of the pack of kits. Advice will be provided on the correct use and interpretation of the HIVST, the need for post-test confirmatory testing in a health facility and the availability of HIV prevention methods including PrEP.

iii. The distributor will be asked to give the test kits to the intended recipients within a seven-day period.

iv. After seven days the helpdesk will contact the distributor and the intended recipients to ascertain whether kits have been received and used, to collect behavioural HIV risk data for the recipients and encourage attendance at a healthcare facility for a confirmatory test. If they have not yet distributed the test kits, the helpline will follow-up at regular intervals to see if distribution has happened. HIVST recipients will be invited to complete the informed consent over the telephone and be enrolled in the study. Follow-up calls will be made to these individuals if necessary. Recipients will be encouraged to consider becoming distributors and advised on the location of community facilities (shops, pharmacies, hairdressers etc.) from where they can obtain the HIVST packs for distribution. This method of HIVST distribution through community-based hubs has been proven to be successful in studies in other Sub-Saharan African settings. [48] A small incentive of USD1:00 will be transferred electronically to the initial distributor for each kit successfully distributed. Successful distribution to peers is defined as the peer having received the HIVST and has been successfully contacted by the helpline to confirm receipt of the HIVST but does not have to use the HIVST or agree to enrol in the study as a distributor. Names and cell numbers will be collected for intended recipients by the study team and stored confidentially.

v. If the recipient chooses to become a distributor, they will go to the community facility and the owner will check using a real-time database that they are eligible. If they pass this screening, they will be given a pack of three HIVST kits for within cluster distribution. If distributors successfully distribute all three HIVST kits within their clusters, they will have the option to collect a further three HIVST kits (up to a total maximum of six HIVST kits) from the community facility. A small remuneration of USD1:00 will be paid to the facility owner for each pack of kits distributed.

vi. After seven days the helpdesk will contact the second level recipients and steps iv) and v) will be repeated until all kits allocated to a particular community have been distributed.

vii. When participants attend a clinic for confirmatory testing, they will return the referral form which was enclosed with the HIVST kit which has a unique barcode and based on their self-reported HIVST result (unreactive/reactive) be screened for PrEP or ART. The outcome of the screening will be recorded in a tick-box on the label and the packaging deposited in a secure box at the clinic from where it will be collected by the study team.

viii. Referral forms, HIVST kits and HIVST packaging will be returned to the central data processing facility for data entry and an additional USD1:00 remuneration will be paid to each individual attending the clinic and participating in a confirmatory HIV test.

ix. All individuals initiating PrEP or ART will be contacted monthly for six months to provide support and to ascertain whether they are still adhering to/continuing with PrEP/ART.

x. Additionally, we will contact all men who report they are still taking PrEP/ART at the end of the follow-up period in order to obtain a dry blood spot to verify the self-report of adherence. This will be sent for analysis in order to assess the intracellular levels of tenofovir diphosphate (TFV-DP) in red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Resident in study site

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3591 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
HIV pre-exposure prophylaxis (PrEP) initiation | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above initiating PrEP

SECONDARY OUTCOMES:
Antiretroviral Therapy initiation | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above initiating Antiretroviral therapy
Antiretroviral Therapy or HIV pre-exposure prophylaxis (PrEP) initiation | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above initiating Antiretroviral therapy
HIV testing | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above taking an HIV test in the clinic.
Confirmed positive HIV test | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above taking an HIV test in the clinic who are diagnosed HIV positive.
HIV testing after the use of an HIV self test | Up to 6 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above taking an HIV test in the clinic after using an HIV test in the previous three months.
Attendance at first PrEP follow-up visit | Up to 8 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above initiating PrEP who return for their first follow-up visit.
Attendance at first ART follow-up visit | Up to 8 months from the start of HIVST distribution in the local intervention clusters
  A comparison between the intervention and control arms of the proportions of men aged 18 and above initiating ART who return for their first follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tanser, PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- BRTI - Manicaland Centre for Public Health Research, Mutare, Manicaland Province, Zimbabwe

DOCUMENTS (1):
  • Study Protocol (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT06370923/Prot_000.pdf